CLINICAL TRIAL: NCT02558881
Title: Evaluation of a Complementary Action of Recruitment of Patients With a Positive Screening Test and Not Realizing Optical Colonoscopy as Part of Organized Colorectal Cancer Screening
Brief Title: Colon Capsule Versus Virtual Colonoscopy for Colorectal Cancer Screening
Acronym: COCAGI
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-757
Record Dates: First submitted 2015-09-18; First posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Colorectal Cancer
Keywords: screening; colorectal cancer; colon capsule; virtual colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Virtual colonoscopy: With virtual colonoscopy, the patient does not need to be hospitalized for examination, which is usually done without hospitalization. A bowel preparation is necessary. It may vary from site to site, but it generally comprises polyethylene glycol or sodium phosphate. The residual stools are "marked" by ingestion of a radiopaque product to differentiate colic lesions. But no contrast agent is injected intravenously. The patient should be supine and a rectal probe is set up to inject either air or CO2. The vesting period does not exceed thirty seconds apnea, and overall completion time of the examination (patient table) is about 10 minutes.
  Interventions: Procedure: Virtual colonoscopy
- Colon capsule: The colon capsule comprises two cameras located at both ends. Image acquisition is set between four to thirty-five images per second. It begins immediately after ingestion of the capsule which allows recording of esophageal and gastric images. She paused for 2 hours (to save batteries) while crossing the small intestine. It is reactivated in the terminal ileum. The films analysis time is approximately 1 hour, and the capsule remains on average 3 hours in the colon.
  Interventions: Procedure: Colon capsule

INTERVENTIONS:
Procedure: Virtual colonoscopy
  Groups: Virtual colonoscopy
Procedure: Colon capsule
  Groups: Colon capsule

SUMMARY:
France is among the countries with a high incidence of colorectal cancer. The prognosis associated with colorectal cancer is related to the development stage of the disease at diagnosis. Thus, when the cancer is detected and treated at an early stage, the survival rate at 5 years was 90%. It is therefore a major issue of screening is widespread in France since the end of 2008.

This screening is based on a two step strategy: 1) the occult blood in the stool (FOBT) and if positive 2) the realization of an optical colonoscopy examination currently regarded as the evaluation procedure colon reference. But as part of this organized screening, 13% of those with a positive FOBT ultimately refuse to have an optical colonoscopy. Under the refusal, virtual colonoscopy may be proposed as an alternative according to the recommendations of the National Health Authority in 2010. But it has never been assessed as part of organized screening. Similarly another alternative is recently developed colic capsule that benefits of development in recent years of the capsule for the small intestine which has become the gold standard for diagnosis of most diseases of the small intestine (bleeding occult, diagnosis of unknown colitis...).

Therefore the study proposes virtual colonoscopy or colon capsule for people with a positive FOBT as part of organized screening and did not realize optical colonoscopy after the usual procedure and complete recovery. This study aims to answer the question of the place of colic capsule as part of organized screening. An economic component is integrated to assess, in terms of health insurance, the cost associated with these two exams, and compare them to the cost of optical colonoscopy.

The proposed study is an observational study of impact of an alternative screening strategy for colorectal cancer whose primary objective is to compare the rate of acceptance of virtual colonoscopy and colon capsule in patients refusing optical colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a positive FOBT at screening organized colorectal cancer, patients who have not achieved optical colonoscopy and who received the usual procedure and complete recovery

Exclusion Criteria:

* None

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a positive FOBT at screening organized colorectal cancer, patients who have not achieved optical colonoscopy and who received the usual procedure and complete recovery.
Sampling Method: Probability Sample
Enrollment: 664 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Acceptance rate of colonic capsule versus virtual colonoscopy. | A period of three months after sending the letter of invitation to an alternative to optical colonoscopy is left to the person.
  Acceptance is defined by the fact that a person having made an appointment for one of the two exams and he went to the review

SECONDARY OUTCOMES:
Success rate of virtual colonoscopy and colon capsule: full review rate of colonic mucosa. | 6 months
Failure rate of examinations by cause | 6 months
  Percentage of bad colic preparations, percentage against-indications, complication rate, percentage capsules have not been to the end of the colon, percentage of other causes (eg. technical ...)
Diagnostic performance of virtual colonoscopy and colon capsule | 6 months
  Percentage of patients with suspected colorectal neoplastic lesions
Achievement rate of optical colonoscopy if a lesion is found, either by virtual colonoscopy, or by colonic capsule | 6 months
  Percentage of patients who achieve an optical colonoscopy after suspected neoplastic colorectal lesion
Sensitivity of virtual colonoscopy and colonic capsule for the diagnosis of cancer, significant additional colorectal polyps, or other polyps | 6 months
  Significant additional colorectal polyps is at least a polyp 6 mm minimum diameter or more than three polyps of any diameter
Specificity of virtual colonoscopy and colonic capsule for the diagnosis of cancer, significant additional colorectal polyps, or other polyps | 6 months
  Significant additional colorectal polyps is at least a polyp 6 mm minimum diameter or more than three polyps of any diameter
Positive and negative predictive values of virtual colonoscopy and colonic capsule for the diagnosis of cancer, significant additional colorectal polyps, or other polyps | 6 months
  Significant additional colorectal polyps is at least a polyp 6 mm minimum diameter or more than three polyps of any diameter
Percentage of cancers diagnosed through virtual colonoscopy or colonic capsule | 6 months
Additional costs generated by the implementation of a complementary action of screening for patients with a positive FOBT and did not realize optical colonoscopy | 6 months
  The costs taken into account will be the direct medical costs of two exams, as well as non-medical direct costs: 1) Letters of invitation to perform any of the tests, 2) Examination conducted (colon capsule or virtual colonoscopy), 3) Letters of Transmittal results

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PONCHON, Professor, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hopsices Civils de Lyon, Lyon, France

REFERENCES:
- [Derived] Pioche M, Ganne C, Gincul R, De Leusse A, Marsot J, Balique J, Fond A, Bretagnolle M, Henry L, Billaud Y, Malezieux R, Lapalus MG, Chambon-Augoyard C, Del Tedesco E, Scalone O, Montoy JC, Russias B, Detry A, Veniat F, Qiu J, Valette PJ, Taillandier A, Saurin JC, Tomczyk-Ferrero J, Gandilhon C, Vecchiato L, Soler-Michel P, Ponchon T. Colon capsule versus computed tomography colonography for colorectal cancer screening in patients with positive fecal occult blood test who refuse colonoscopy: a randomized trial. Endoscopy. 2018 Aug;50(8):761-769. doi: 10.1055/s-0044-100721. Epub 2018 Feb 27. PMID 29486502